CLINICAL TRIAL: NCT06414551
Title: Characteristics of Calcification in a Chronic Total Occlusion on Computed Tomography Coronary Angiogram and Percutaneous Coronary Intervention Outcomes- a Single Centre Observational Study
Brief Title: Calcification on CTCA of a CTO and PCI Outcomes
Status: Recruiting | Type: Observational
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Vinoda Sharma, Cardiology Specialty Lead, Honorary Associate Professor, Interventional Cardiologist, Sandwell & West Birmingham Hospitals NHS Trust
Other Study IDs: IRAS Project ID: 333718
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Calcification; Computed Tomography Angiography
Keywords: CTCA; CTO
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CTO patients who underwent attempted PCI: Patients with coronary CTO who underwent attempt at PCI and also underwent a CTCA

SUMMARY:
A chronic total occlusion (CTO) is present in 15-20% of patients who are referred for invasive coronary angiography. CTO Percutaneous Coronary Intervention (PCI) procedure success rates have increased over the years and can be as high as 90% when performed by high-volume CTO operators.Procedurally, excess calcification in the CTO anatomy is one factor which makes it difficult to complete the procedure or obtain ideal stent expansion. Excess calcification is best identified by Computed Tomography Coronary Angiography (CTCA) rather than invasive angiography.

The investigators plan to retrospectively evaluate CTCA in patients who underwent CTO PCI and correlate calcification characteristics with CTO PCI outcomes and tools utilised for calcium modification.

DETAILED DESCRIPTION:
Cohort: All coronary CTO patients who underwent a PCI attempt and also underwent CTCA at our centre in the last 5 years.

Method of identifying and consenting patients: Screening of our local database to identify suitable patients who fulfil the inclusion/exclusion criteria. These patients will be telephoned and the consent form and participant information sheet will be maile dot them along with a self addressed stamped envelope.On receipt of the consent form, we will countersign it and return a copy to the patient. Consented patients' images and reports of the CTCA and CTO PCI will be reviewed.

Characteristics of calcification in the CTO on the CTCA will be evaluated including site, density and quantity of calcification. This will be correlated with CTO PCI outcomes of success and failure. Also this will be correlated with use of calcium modification tools for the CTO PCI.

* Baseline and demographic as well as procedural data will be compared with CTO PCI outcomes and presence/characteristics of calcification.
* Characteristics of calcification in the CTO assessed will include: site, density in Hounsfield units and quantity.
* Site of calcification (proximal, body or distal) will be correlated with the CTO PCI outcome by chi square analysis.
* Calcium density (in Hounsfield Units) on the CTCA will be correlated with successful versus failed CTO PCI by ROC curve analysis.
* Quantity of calcification will be assessed as a percentage of the cross section of the CTO body (as <50%, 50-75% and 75-100%) and correlated with CTO PCI success by contingency analysis.
* Use of calcium modification tools will be correlated with CTO PCI outcome (success or failure) and density of calcification on CTCA (ROC curve and ANOVA).
* Categorical variables will be compared by the chi square or Fisher's test and continuous variables will be compared by the Mann Whitney U test. In addition, based on CTO PCI outcome of success or failure, patients will be compared for demographics and procedural variables.
* Categorical variables will be presented as percentage and compared with the chi square or Fisher's test
* Continuous variables will be presented as median (range) and compared with student's t-test or Mann Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting all the below criteria will be included

  * ≥18 years
  * Previous CTO PCI attempt in the last 5 years
  * Undergone CTCA either pre or post CTO PCI
  * Adequate CTCA images for analysis

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded

  * <18 years of age
  * Did not undergo CTCA
  * Inadequate/degraded CTCA images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary CTO who underwent attempt at PCI and also underwent CTCA
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of characteristics of calcification with CTO PCI outcome (success or failure) | up to 24 hours
  Success or failure

SECONDARY OUTCOMES:
Utility of calcium modifying tools for the CTO PCI procedure and correlation with severity of calcification | up to 24 hours
  Percentage of patients in whom any calcium modifying tool was used and the corelation of this with the severity of calcification.

CONTACTS AND LOCATIONS:
Overall Officials: Vinoda Sharma, FRCP, Principal Investigator — Sandwell & West Birmingham Hospitals NHS Trust
Locations (1):
- Birmingham City Hospital, Sandwell and West Birmingham NHS Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tajti P, Brilakis ES. Chronic Total Occlusion Percutaneous Coronary Intervention: Evidence and Controversies. J Am Heart Assoc. 2018 Jan 12;7(2):e006732. doi: 10.1161/JAHA.117.006732. No abstract available. PMID 29330258
- [Background] Patel VG, Brayton KM, Tamayo A, Mogabgab O, Michael TT, Lo N, Alomar M, Shorrock D, Cipher D, Abdullah S, Banerjee S, Brilakis ES. Angiographic success and procedural complications in patients undergoing percutaneous coronary chronic total occlusion interventions: a weighted meta-analysis of 18,061 patients from 65 studies. JACC Cardiovasc Interv. 2013 Feb;6(2):128-36. doi: 10.1016/j.jcin.2012.10.011. Epub 2013 Jan 23. PMID 23352817
- [Background] Sharma V, Jadhav ST, Harcombe AA, Kelly PA, Mozid A, Bagnall A, Richardson J, Egred M, McEntegart M, Shaukat A, Oldroyd K, Vishwanathan G, Rana O, Talwar S, McPherson M, Strange JW, Hanratty CG, Walsh SJ, Spratt JC, Smith WH. Impact of proctoring on success rates for percutaneous revascularisation of coronary chronic total occlusions. Open Heart. 2015 Mar 28;2(1):e000228. doi: 10.1136/openhrt-2014-000228. eCollection 2015. PMID 25852949
- [Background] Simon W. The Consistent CTO Study. 2018.
- [Background] Gada H, Whitlow PL, Marwick TH. Establishing the cost-effectiveness of percutaneous coronary intervention for chronic total occlusion in stable angina: a decision-analytic model. Heart. 2012 Dec;98(24):1790-7. doi: 10.1136/heartjnl-2012-302581. Epub 2012 Oct 4. PMID 23038791
- [Background] Grantham JA, Jones PG, Cannon L, Spertus JA. Quantifying the early health status benefits of successful chronic total occlusion recanalization: Results from the FlowCardia's Approach to Chronic Total Occlusion Recanalization (FACTOR) Trial. Circ Cardiovasc Qual Outcomes. 2010 May;3(3):284-90. doi: 10.1161/CIRCOUTCOMES.108.825760. Epub 2010 Apr 13. PMID 20388873
- [Background] Olivari Z, Rubartelli P, Piscione F, Ettori F, Fontanelli A, Salemme L, Giachero C, Di Mario C, Gabrielli G, Spedicato L, Bedogni F; TOAST-GISE Investigators. Immediate results and one-year clinical outcome after percutaneous coronary interventions in chronic total occlusions: data from a multicenter, prospective, observational study (TOAST-GISE). J Am Coll Cardiol. 2003 May 21;41(10):1672-8. doi: 10.1016/s0735-1097(03)00312-7. PMID 12767645
- [Background] Werner GS, Martin-Yuste V, Hildick-Smith D, Boudou N, Sianos G, Gelev V, Rumoroso JR, Erglis A, Christiansen EH, Escaned J, di Mario C, Hovasse T, Teruel L, Bufe A, Lauer B, Bogaerts K, Goicolea J, Spratt JC, Gershlick AH, Galassi AR, Louvard Y; EUROCTO trial investigators. A randomized multicentre trial to compare revascularization with optimal medical therapy for the treatment of chronic total coronary occlusions. Eur Heart J. 2018 Jul 7;39(26):2484-2493. doi: 10.1093/eurheartj/ehy220. PMID 29722796
- [Background] Mashayekhi KA, Pyxaras SA, Werner GS, Galassi AR, Garbo R, Boudou N, Leibundgut G, Avran A, Bryniarski L, Bufe A, Sianos G, Di Mario C. Contemporary issues of percutaneous coronary intervention in heavily calcified chronic total occlusions: an expert review from the European CTO Club. EuroIntervention. 2023 Jun 5;19(2):e113-e122. doi: 10.4244/EIJ-D-22-01096. PMID 36971414
- [Background] Morino Y, Abe M, Morimoto T, Kimura T, Hayashi Y, Muramatsu T, Ochiai M, Noguchi Y, Kato K, Shibata Y, Hiasa Y, Doi O, Yamashita T, Hinohara T, Tanaka H, Mitsudo K; J-CTO Registry Investigators. Predicting successful guidewire crossing through chronic total occlusion of native coronary lesions within 30 minutes: the J-CTO (Multicenter CTO Registry in Japan) score as a difficulty grading and time assessment tool. JACC Cardiovasc Interv. 2011 Feb;4(2):213-21. doi: 10.1016/j.jcin.2010.09.024. PMID 21349461
- [Background] Christopoulos G, Kandzari DE, Yeh RW, Jaffer FA, Karmpaliotis D, Wyman MR, Alaswad K, Lombardi W, Grantham JA, Moses J, Christakopoulos G, Tarar MNJ, Rangan BV, Lembo N, Garcia S, Cipher D, Thompson CA, Banerjee S, Brilakis ES. Development and Validation of a Novel Scoring System for Predicting Technical Success of Chronic Total Occlusion Percutaneous Coronary Interventions: The PROGRESS CTO (Prospective Global Registry for the Study of Chronic Total Occlusion Intervention) Score. JACC Cardiovasc Interv. 2016 Jan 11;9(1):1-9. doi: 10.1016/j.jcin.2015.09.022. PMID 26762904
- [Background] Maeremans J, Spratt JC, Knaapen P, Walsh S, Agostoni P, Wilson W, Avran A, Faurie B, Bressollette E, Kayaert P, Bagnall AJ, Smith D, McEntegart MB, Smith WHT, Kelly P, Irving J, Smith EJ, Strange JW, Dens J. Towards a contemporary, comprehensive scoring system for determining technical outcomes of hybrid percutaneous chronic total occlusion treatment: The RECHARGE score. Catheter Cardiovasc Interv. 2018 Feb 1;91(2):192-202. doi: 10.1002/ccd.27092. Epub 2017 May 4. PMID 28471074
- [Background] Szijgyarto Z, Rampat R, Werner GS, Ho C, Reifart N, Lefevre T, Louvard Y, Avran A, Kambis M, Buettner HJ, Di Mario C, Gershlick A, Escaned J, Sianos G, Galassi A, Garbo R, Goktekin O, Meyer-Gessner M, Lauer B, Elhadad S, Bufe A, Boudou N, Sievert H, Martin-Yuste V, Thuesen L, Erglis A, Christiansen E, Spratt J, Bryniarski L, Clayton T, Hildick-Smith D. Derivation and Validation of a Chronic Total Coronary Occlusion Intervention Procedural Success Score From the 20,000-Patient EuroCTO Registry: The EuroCTO (CASTLE) Score. JACC Cardiovasc Interv. 2019 Feb 25;12(4):335-342. doi: 10.1016/j.jcin.2018.11.020. Epub 2019 Jan 30. PMID 30711551
- [Background] Opolski MP, Achenbach S, Schuhback A, Rolf A, Mollmann H, Nef H, Rixe J, Renker M, Witkowski A, Kepka C, Walther C, Schlundt C, Debski A, Jakubczyk M, Hamm CW. Coronary computed tomographic prediction rule for time-efficient guidewire crossing through chronic total occlusion: insights from the CT-RECTOR multicenter registry (Computed Tomography Registry of Chronic Total Occlusion Revascularization). JACC Cardiovasc Interv. 2015 Feb;8(2):257-267. doi: 10.1016/j.jcin.2014.07.031. PMID 25700748
- [Background] Panuccio G, Skurk C, Landmesser U, Abdelwahed YS. Double "full moon" CTO plaque detected by computed tomography could predict high-grade debulking techniques: A case-report. Clin Case Rep. 2023 May 18;11(5):e7325. doi: 10.1002/ccr3.7325. eCollection 2023 May. PMID 37215968
- [Background] Improvement N. 2019/20 National Tariff Payment System. In: system Ntp, editor. 2019.